CLINICAL TRIAL: NCT01797614
Title: Measuring the Change of Intra-abdominal Pressures of the Intensive Care Unit Patients During the Spontaneous Breathing Trial
Brief Title: Intra-abdominal Pressures During the Spontaneous Breathing Trial
Acronym: IAP_SBT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201108062RC
Record Dates: First submitted 2013-02-20; First posted 2013-02-22 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Respiratory Failure
Keywords: intra-abdominal pressure; spontaneous breathing trail; weaning
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Increased intra-abdominal pressure (IAP) affects pulmonary dynamics. However, little is studied whether pulmonary dynamics affects IAP. We hypothesize that the change of IAP can also reflect the change of pulmonary dynamics. In this study, we choose patients who received spontaneous breathing trial to answer the hypothesis.

DETAILED DESCRIPTION:
During the weaning process, we tapered down the respiratory support from mechanical ventilation and recruited respiratory muscles to work. Previous study showed that transdiaphragmatic pressure was increasing while pressure support was reducing. However, the transdiaphragmatic pressure required invasive procedure to measure and not used frequently in weaning. IAP reflects the pleural pressure. If the PEEP is not changed, change of IAP is largely due to change of transpulmonary pressure.

Study Aim:

1. To evaluate the patterns of change of IAP during SBT
2. To predict success of SBT by the change of IAP
3. To predict weaning outcome by the change of IAP

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with endotracheal intubation in the intensive care unit
* The clinical condition is considered to prepare for weaning assessment

Exclusion Criteria:

* tracheostomy
* severe heart failure, heart disease or arrhythmia
* upper airway obstruction related respiratory failure
* poor cooperation due to agitation
* no foley catheter in place or had been removed
* baseline IAP above 20 mmHg

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with endotracheal intubation and are preparing for weaning assessment
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-07 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the patterns of change of IAP during SBT | 30min, 60min, 120min
  30min, 60min, 120min during a 2-hr SBT

SECONDARY OUTCOMES:
To predict success of SBT by the change of IAP | 0 min, 30 min, 120 min
  To predict success of 2-hour IAP the change of IAP between 0 min and 30 min, and tha change of IAP beween 0 min and 120 min
To predict weaning success by the change of IAP | 0 min, 30 min, 120 min
  To predict weaning success by the change of IAP between 0 min and 30 min, and tha change of IAP beween 0 min and 120 min

CONTACTS AND LOCATIONS:
Overall Officials: Nin-Chieh Hsu, MD, Principal Investigator — National Taiwan University Hospital
Locations (2):
- Taiwan (2):
  - Nin-Chieh Hsu, Taipei, Taipei
  - National Taiwan University Hospital, Taipei